CLINICAL TRIAL: NCT01311479
Title: Osteopathic Manipulation as a Therapeutic Intervention for Female Interstitial Cystitis Patients With Sacroiliac Joint Dysfunction
Brief Title: Osteopathic Manipulation for Female Interstitial Cystitis Patients With Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pelvic and Sexual Health Institute (Other)
Collaborators: Interstitial Cystitis Association (ICA) (Other)
Responsible Party: Principal Investigator, Kristene Whitmore, M.D., Medical Director, Pelvic and Sexual Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMT-09
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Interstitial Cystitis; Sacroiliac Joint Somatic Dysfunction
Keywords: Osteopathic Manipulation; Interstitial Cystitis; Sacroiliac Joint Dysfunction
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic Manipulation (Active Comparator): Patients will be evaluated and examined by an Osteopathic physician. This examination will consist of full osteopathic structural exam, and a focused examination of the sacroiliac joint and the surrounding musculature.
  Subjects will then be treated based on the objective findings of the examination. Since the structural exam includes the whole body, other structural abnormalities will likely be identified and possible require treatment to aid in treatment of SIJ. Subjects will also be taught stretching routines in order to aid in treatment of the dysfunction.
  Interventions: Procedure: Osteopathic Manipulation Therapy
- Massage Therapy (Active Comparator): Our control group will receive the same structural exam, and focused examination. Their treatment will involve massage, in an area not associated with the musculature of the SIJ. This will serve to identify a possible placebo effect, associated with simply providing a healing touch without focused treatment.
  Interventions: Procedure: Osteopathic Manipulation Therapy

INTERVENTIONS:
Procedure: Osteopathic Manipulation Therapy — Subjects will then be treated based on the objective findings of the examination. Since the structural exam includes the whole body, other structural abnormalities will likely be identified and possible require treatment to aid in treatment of SIJ. Subjects will also be taught stretching routines in order to aid in treatment of the dysfunction.
  Our control group will receive the same structural exam, and focused examination. Their treatment will involve massage, in an area not associated with the musculature of the SIJ. This will serve to identify a possible placebo effect, associated with simply providing a healing touch without focused treatment.

SUMMARY:
The proposed study will evaluate the effectiveness of Osteopathic manipulation of the sacro-iliac joint (SIJ) and the lumbar spine in symptomatic female interstitial cystitis (IC) patients with sacro-iliac joint dysfunction.

It is predicted that Osteopathic manipulation for a period of 12 weeks will result in subjective indices of increased comfort and objective indices of lower O'Leary-Sant Questionnaire, Pelvic Floor Impact Questionnaire (PIFQ-7), Female Sexual Function Index (FSFI) and SF-12 scores, lower visual analog scores for pain and urgency, decreased frequency on voiding diary and greater variation in resting/contraction perineometry scores.

DETAILED DESCRIPTION:
Patients will be evaluated and examined by an Osteopathic physician. This examination will consist of full osteopathic structural exam, and a focused examination of the sacroiliac joint and the surrounding musculature.

Subjects will then be treated based on the objective findings of the examination. Since the structural exam includes the whole body, other structural abnormalities will likely be identified and possible require treatment to aid in treatment of SIJD. Subjects will also be taught stretching routines in order to aid in treatment of the dysfunction.

Our control group will receive the same structural exam, and focused examination. Their treatment will involve massage, in an area not associated with the musculature of the SIJ. This will serve to identify a possible placebo effect, associated with simply providing a healing touch without focused treatment.

All of the subjects will be evaluated with standardized IC questionnaires at time of initial visit and subsequently re-evaluated with the same questionnaire in 4 week intervals. The patients will be followed for up to 6 months after treatment and evaluated at this time.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 18 years of age
* Patients who have osteopathic dysfunction
* Patients with the Diagnosis of IC and Sacroiliac joint dysfunction
* Patients currently stable on or off of a treatment regimen for IC for the past one month
* Patients not currently undergoing physical therapy for pelvic floor dysfunction or SI joint dysfunction
* Patients who have not used narcotics, skeletal muscle relaxants, or bladder instillations for the past month
* Willingness to participate in the trial by signing an informed consent

Exclusion Criteria:

* Pregnancy
* Pelvic Masses
* Patients with an Interstim neuromodulator implant
* Patients requiring narcotics, bladder instillations, or skeletal muscle relaxants
* History of vaginal or abdominal pelvic surgery within the last 3 months
* Having a bladder over-distention within the last 1 month
* Malignancy
* Known spinal arthropathies
* Hip replacements or other surgical stabilization
* Herniated disks
* Spinal stenosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in Scores of Validated questionnaires pertaining to Interstitial Cystitis problems and symptoms | Biweekly for three months
  It is predicted that Osteopathic manipulation for a period of 12 weeks will result in subjective indices of increased comfort and objective indices of lower O'Leary-Sant Questionnaire, Pelvic Floor Impact Questionnaire (PIFQ-7), Female Sexual Function Index (FSFI) and SF-12 scores, lower visual analog scores for pain and urgency, decreased frequency on voiding diary and greater variation in resting/contraction perineometry scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kristene E Whitmore, M.D., Principal Investigator — Pelvic and Sexual Health Institute
Locations (1):
- Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania, United States